CLINICAL TRIAL: NCT03749018
Title: A Phase II Study of Nivolumab in Combination With DA-REPOCH Followed by Short Course Nivolumab Consolidation in Patients With Aggressive B-Cell Non-Hodgkin's Lymphoma
Brief Title: Nivolumab With DA-REPOCH Chemotherapy Regimen in Treating Patients With Aggressive B-Cell Non-Hodgkin's Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: David Bond, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, David Bond, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-18281; NCI-2018-02699 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Aggressive Non-Hodgkin Lymphoma; Ann Arbor Stage I Primary Mediastinal (Thymic) Large B-Cell Cell Lymphoma; Ann Arbor Stage II B-Cell Non-Hodgkin Lymphoma; Ann Arbor Stage II Primary Mediastinal (Thymic) Large B-Cell Cell Lymphoma; Ann Arbor Stage III B-Cell Non-Hodgkin Lymphoma; Ann Arbor Stage III Primary Mediastinal (Thymic) Large B-Cell Cell Lymphoma; Ann Arbor Stage IV B-Cell Non-Hodgkin Lymphoma; Ann Arbor Stage IV Primary Mediastinal (Thymic) Large B-Cell Cell Lymphoma; Diffuse Large B-Cell Lymphoma; High Grade B-Cell Lymphoma With MYC and BCL2 and/or BCL6 Rearrangements; High Grade B-Cell Lymphoma, Not Otherwise Specified; Indolent Non-Hodgkin Lymphoma; Mediastinal B-Cell Lymphoma, Unclassifiable, With Features Intermediate Between Diffuse Large B-Cell Lymphoma and Classic Hodgkin Lymphoma; Transformed Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Doxorubicin; Etoposide; Nivolumab; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, DA-REPOCH) (Experimental): Patients receive rituximab IV and nivolumab IV over 60 minutes on day 1. Patients also receive etoposide, vincristine sulfate and doxorubicin hydrochloride IV continuously over 96 hours, cyclophosphamide IV bolus, and prednisone PO on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. After course 6, patients receive nivolumab IV over 60 minutes on day 1 every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Biological: Nivolumab; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Drug: Vincristine Sulfate — Give IV
  Other Names: Kyocristine; Leurocristine sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies how well nivolumab works with the DA-REPOCH chemotherapy regimen in treating patients with aggressive B-cell non-Hodgkin lymphoma. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body?s immune system attack the cancer, and may interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as dose-adjusted rituximab, etoposide, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin hydrochloride (DA-REPOCH), work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving nivolumab with DA-REPOCH may work better in treating patients with aggressive B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine 2-year progression-free survival (PFS) of nivolumab in combination with DA-REPOCH with short course nivolumab maintenance.

SECONDARY OBJECTIVES:

I. To determine the objective response rate (ORR), complete response (CR) rate, and duration of response to nivolumab in combination with DA REPOCH with short course nivolumab maintenance.

II. To establish that nivolumab in combination with DA-REPOCH with short course nivolumab maintenance is feasible at standard dosing.

III. To establish the toxicity profile of nivolumab in combination with DA-REPOCH with short course nivolumab maintenance at standard dosing.

EXPLORATORY OBJECTIVES:

I. To correlate the presence of major histocompatibility complex (MHC) class I and II by immunohistochemistry (IHC) with PFS.

II. To correlate tumor and microenvironment expression of PD-L1 and microenvironment expression of PD-1 with PFS.

III. To correlate cell of origin, MYC and Bcl-2 expression, Epstein-Barr virus (EBV)-positivity, and Ki67 proliferation index with response to treatment.

IV. To determine the effect of nivolumab in combination with DA-REPOCH on immune cell subsets in the peripheral blood over time.

V. To correlate circulating tumor (ct) deoxyribonucleic acid (DNA) with disease response by positron emission tomography (PET) imaging.

VI. To track clonal evolution and detect the emergence of treatment-resistance by ct-DNA monitoring.

OUTLINE:

Patients receive rituximab intravenously (IV) and nivolumab IV over 60 minutes on day 1. Patients also receive etoposide, vincristine sulfate and doxorubicin hydrochloride IV continuously over 96 hours, cyclophosphamide IV bolus, and prednisone orally (PO) on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. After course 6, patients receive nivolumab IV over 60 minutes on day 1 every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 3 years, and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Measurable disease (defined as >= 1.5 cm in diameter) or at least one PET avid area of disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Absolute neutrophil count (ANC) >= 1,000 /mcL (within 16 days of treatment initiation).
* Platelets >= 75,000 / mcL in the absence of transfusion support within 7 days of determining eligibility (within 16 days of treatment initiation).
* Hemoglobin >= 8 g/dL (within 16 days of treatment initiation).
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance >= 40 mL/min creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) (within 16 days of treatment initiation).

  * Creatinine clearance should be calculated per institutional standard.
* Serum total bilirubin =< 1.5 X ULN OR except subjects with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL (within 16 days of treatment initiation).
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 X ULN (within 16 days of treatment initiation).
* Female subject of childbearing potential should have a negative serum pregnancy at screening.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 5 months following the last dose of nivolumab. Subjects should agree to ongoing pregnancy testing during the course of the study and after the end of study therapy. Female subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 7 months following the last dose of nivolumab. Males must refrain from donating sperm during study participation and for 7 months after the last dose of nivolumab.
* Revised Ann Arbor stage II-IV disease

  * Stage I primary mediastinal B-cell lymphoma or mediastinal B cell lymphoma unclassifiable with features intermediate between DLBCL and classical Hodgkin?s lymphoma will also be eligible.
* Be willing and able to understand and give written informed consent and comply with all study related procedures.

Exclusion Criteria:

* Known hypersensitivity to any of the study drugs.
* History of other malignancy that could affect compliance with the protocol or interpretation of the results.
* Has a diagnosis of immunodeficiency excluding human immunodeficiency virus (HIV) infection or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Subjects may use topical or inhaled corticosteroids or low-dose steroids (=< 10 mg of prednisone or equivalent per day) as therapy for comorbid conditions. During study participation, subjects may receive systemic or enteric corticosteroids as needed for treatment-emergent comorbid conditions.
* Has a known history of active TB (Bacillus tuberculosis).
* Prior systemic chemotherapy for lymphoma with the exception of corticosteroids for palliation of symptoms and patients with prior indolent non-Hodgkin lymphoma (NHL) treated with single agent rituximab.
* Has known active central nervous system (CNS) lymphoma.
* Richter?s transformation from chronic lymphocytic leukemia (CLL).
* Major surgery within 3 weeks prior to start of study treatment.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Conditions expected to not recur in the absence of an external trigger.
* Has an active infection requiring intravenous systemic therapy or uncontrolled systemic infection including viral, bacterial, or fungal.
* Is unable to swallow capsules or malabsorption syndrome, disease or condition significantly affecting gastrointestinal function.
* Clinically significant cardiovascular disease, including uncontrolled arrhythmia, New York Association class 2- 4 congestive heart failure, or history of myocardial infarction within 6 months.
* Known contraindication to any medication in the treatment plan, including clinically significant peripheral neuropathy.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Female patients who are not surgically sterile or postmenopausal (for at least 1 year) must practice at least one of the following methods of birth control throughout the duration of study participation and for at least 5 months after study treatment:

  * Total abstinence from hetero-sexual intercourse
  * A vasectomized partner
  * Hormonal contraceptives (oral, parenteral, vaginal ring, or transdermal) that started at least 3 months prior to study drug administration
  * Double-barrier method (condom + diaphragm or cervical cup with spermicidal contraceptive sponge, jellies, or cream)
  * Non-vasectomized male patients must comply with at least one of the following methods of birth control throughout the duration of study participation and for at least 3 months after study treatment:
  * A partner who is surgically sterile or postmenopausal (for at least 1 year) or who is taking hormonal contraceptives (oral, parenteral, vaginal ring, or transdermal) for at least 3 months prior to study drug administration
  * Total abstinence from hetero-sexual intercourse
  * Double-barrier method (condom + diaphragm or cervical cup with spermicidal, contraceptive sponge, jellies, or cream).
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Acute hepatitis C (defined as positive hepatitis C virus (HCV) ribonucleic acid (RNA) [qualitative] and diagnosis within the past 6 months).
* Positive hepatitis C antibody with evidence of cirrhosis.
* Active hepatitis B (subjects with a positive hepatitis B virus [HBV] core antibody or surface antigen are eligible as long as they have an undetectable HBV DNA polymerase chain reaction [PCR] and receive concurrent antiviral therapy with entecavir or tenofovir, and continued for a minimum of 6 months after completion of therapy).
* HIV infection AND CD4 count < 100 cells/ mm^3, evidence of resistant strain of HIV, or HIV viral load >= 50 copies HIV RNA/mL if on highly active antiretroviral therapy (HAART) or HIV viral load >= 10,000 copies HIV RNA/mL if not on anti-HIV therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2026-02-02 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From start of treatment to progression or death, whichever occurs first, assessed at 2 years
  Will be estimated by the method of Kaplan-Meier and the estimate will be provided with 95% confidence intervals. Depending on the number of events, Cox regression model may be used to explore the association between baseline clinical variables and PFS in a univariable manner.

SECONDARY OUTCOMES:
Objective response rate | Up to 8 years
  Will be calculated with patients who achieve complete response (CR) or partial response (PR) at end of induction therapy as the numerator and all eligible patients who start treatment as the denominator, with a 95% binomial confidence interval provided. CR rate will be analyzed in the same way.
Duration of response defined for all patients who have achieved an objective response (CR or PR) | From date of which patient?s response is documented to the date of progression or death, censoring event-free patients at the time of last follow-up, assessed up to 8 years
  Will be described using the method of Kaplan-Meier.
Incidence of adverse events per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | Up to 30 days post-treatment
  All adverse events will be summarized and tabulated across all patients who received any treatment with a focus on severe (grade 3+) adverse events and toxicities that are deemed at least possibly related to study treatment.

OTHER OUTCOMES:
Major histocompatibility complex (MCH) class I and II expression | Up to 8 years
  Will be correlated with PFS and be explored using graphical methods such as Kaplan-Meier curves.
Expression of PD-1 and PD-L1 with PFS | Up to 8 years
  Will be correlated with PFS and explored using graphical methods such as Kaplan-Meier curves.
Somatic mutations detection by circulating tumor (ct)-deoxyribonucleic acid (DNA) over time | Up to 8 years
  Will be described using either box plots or individual time plots grouped by relevant subcategories (e.g. response) to help identify potential patterns. Wilcoxon signed rank test will be used to compare baseline expression with values measured at time of relapse.

CONTACTS AND LOCATIONS:
Overall Officials: David A Bond, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu